CLINICAL TRIAL: NCT03802383
Title: A Study on the Relationship Between the Trans-diaphragmatic Pressure and the Contraction of the Diaphragm
Brief Title: The Relationship Between Trans-diaphragmatic Pressure and Diaphragmatic Contraction
Status: Recruiting | Type: Observational
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, DEMOSTHENES MAKRIS, Associate Professor of Critical Care Medicine, University of Thessaly
Other Study IDs: 3531/29.06.2018
Record Dates: First submitted 2018-12-22; First posted 2019-01-14 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Weaning Failure; Respiratory Paralysis; Respiratory Failure
MeSH Terms: conditions — Respiratory Paralysis; Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Through this study the investigators aim to clarify the relationship between trans-diaphragmatic pressure and various parameters of the diaphragmatic contraction evaluated by ultrasound. Moreover, a lung ultrasound exam will be performed at the end of spontaneous breathing, resistive breathing and maximal inspiratory pressure maneuver (MIP) in order to assess with the use of B-lines for extravascular lung water (EVLW). The following parameters will be studied: esophageal pressure, gastric pressure, diaphragm thickness at peak inspiration (Tdi,pi), diaphragm thickness at end expiration (Tdi,ee), diaphragm thickening (Tdi,pi - Tdi,ee), diaphragm thickness fraction [TFdi=(Tdi,pi - Tdi,ee)/Tdi,ee], diaphragm excursion (Dec), Maximal Inspiratory pressure (M.I.P), Pressure-Time product of the esophageal pressure (PΤPes),Tension Time Diaphragm Index (T.T.Di) and the rapid shallow breathing index (R.S.B.I.). These measurements will be made in two phases.Firstly, during the spontaneous breathing trial and secondly during spontaneous breathing through an airway of reduced diameter.Furthermore, during the M.I.P. test the aforementioned ultrasound parameters will be measured. The aim of this study is to discover new means of a successful prediction of weaning in the first 48 hours following extubation.

DETAILED DESCRIPTION:
Protocol

The patients will enter a Spontaneous Breathing Trial (S.B.T.) for sixty minutes. During the S.B.T. the desirable measurements will be made: transdiaphragmatic pressure, diaphragm thickening, Tdi,pi , Tdi,ee , TFdi, Di,e, Maximal Inspiratory Pressure (M.I.P.) , Rapid Shallow Breathing Index (R.S.B.I.). If the S.B.T. is successful then the patient will be removed from the mechanical ventilator. For the next 48 hours the patient will be monitored for distress signs and thus be reintubated or if the weaning of the patient was successful extubation.

Flow chart of the study

1. The patient meets the S.B.T. criteria.
2. The patient is placed in a semi recumbent position.
3. A nasogastric tube attached with two balloons, which are connected with a pressure transducer, one placed in the stomach and the other one in the lower third of the esophagus.
4. The balloons will be connected with a Hans Rudolph pneumotachograph for the measurement of the tidal volume, the flow and the esophageal pressure.
5. An occlusion test will be performed to make sure the esophageal balloon is correctly placed.
6. Measurement of Pes, Pgas and simultaneous sonographic measurements (Diaphragm thickening, Tdipi, Tdiee, Dex, TFdi) during the S.B.T. with the patient being in t-tube.
7. Performance of a MIP maneuver.
8. Measurement of the same parameters during an S.B.T. with an airway of reduced diameter (resistive breathing).
9. Performance of lung ultrasound for B-lines estimation at the end of SBT, MIP and the resistive breathing)
10. If the S.B.T. is successful according to the R.S.B.I. the patient will be disconnected from the mechanical ventilation.
11. Monitoring of the patient for the next 48 hours, for the extubation respiratory distress syndrome or reintubation for another reason.
12. Further monitoring for 30 days in order to measure the time spent in mechanical ventilation

Definitions

Transdiaphragmatic pressure

Pdi will be measured with the use of a nasogastric catheter which has 2 balloons attached at 25 cm and 10 cm from it's distal end. The balloons, of 7 cm length, will be connected with a pressure transducer and with the use of a linear pneumotachometer Hans Rudolph RSS 100HR the graphic representation of the pressures will be displayed in a computer monitor. The balloons will contain 0,5-1 ml of air and will be placed in the stomach and the lower third of the esophagus. To ensure the correct positioning of the balloons an occlusion test (Baydur test) will be performed ,where the similar fluctuations between the esophageal and the airway pressure will be affirmative. As long as the stomach balloon is concerned the positive pressures during the inspiration will be affirmative of the correct positioning.

Tension Time Diaphragm Index

Ttdi is used as an index of diaphragmatic exhaustion. Measurements above 0,15 are indicative of the diaphragmatic incapability to maintain spontaneous breathing for more than 45 minutes, whence the naming of Ttdi critical

Ttdi = (Pdi/Pdi,max)x(TixTtot)

Rapid Shallow Breathing Index

Rapid Shallow Breathing Index (R.S.B.I.) is a method used for predicting the weaning outcome. It is measured during spontaneous breathing and equates to the ratio of respiratory rate per minute (RR) to the tidal volume (Vt) expressed in liters.

R.S.B.I. = RR/Vt

It has been shown that an R.S.B.I. values below 105 breaths/min/L can predict a successful weaning.

Maximal Inspiratory Pressure

Maximal Inspiratory Pressure (M.I.P.) is used as a predictive factor of the weaning outcome. It is measured with a manometer placed in a fully occluded airway, while the patient tries to breathe through it for 20 seconds. The highest pressure value is named M.I.P. It has been shown that values below -25 cmH2O are indicative of a positive weaning outcome.

Pressure-Time Product of the Esophageal pressure

PTPes was calculated as the area enclosed within the Pes trace, the superimposed recoil of the chest wall and onset and end of inspiratory flow. The chest wall recoil pressure was calculated as 4% of predicted vital capacity.

Diaphragm Ultrasound

The diaphragmatic function is assessed during spontaneous breathing and during breathing with an airway of reduced diameter. The diaphragmatic movement is assessed with ultrasound (Phillips iE33) using a Linear 3-11 MHz head. The ultrasound probe is placed in the mid axillary line perpendicular to the zone of apposition between the 8th-10th intercostal spaces. In this position, the diaphragm is shown as a non-echogenic layer between two echogenic layers which represent the diaphragmatic pleura and the abdominal peritoneum. With this technique the diaphragmatic thickening (Tdi,pi - Tdi,ee), diaphragmatic thickness at end-expiration (Tdi,ee) and end-inspiration (Tdi,pi), diaphragmatic excursion Di,e and diaphragmatic thickening fraction TFdi are measured. All the measurements are made using M-Mode Sonography.

Lung Ultrasound

Lung ultrasound (LUS) was performed in the anterior chest to estimate the number of B-Lines at the end of each phase. A restrictive two-region LUS test, conducted in the anterior chest region, was considered to assess EVLW during these maneuvers. Lung ultrasound was conducted at the end of SBT, MIP and RBT to evaluate for the generation of B-lines during each of these phases. Afterwards patients were categorized, according to the number of B-lines present, in four categories depending on the total number of B-lines 0: 0 B-lines, 1: 1-2 B-lines, 2: 3-7 B-lines, 3: >7 B-lines.

ELIGIBILITY:
Inclusion Criteria:

Patients meeting the following standards.

* Respiratory Criteria

  * PaO2≥ 60mmHg with Fraction of Inspired Oxygen (FiO2) ≤ 40-50% & Positive End Expiratory Pressure (PEEP) ≤ 5-8 cm H2O
  * PaCO2 normal or at the level of reference (allowed hypercapnia is allowed)
  * Patient is able to start ventilatory effort
* Cardiovascular Criteria

  * Absence of myocardial ischemia
  * Heart Rate ≤140 bpm
  * Arterial Pressure normal without vasoconstriction or with minimum vasoconstriction support
* Adequate level of consciousness

  o Glasgow Coma Scale (GCS ≥ 13)
* Absence of other reversible comorbidities

  * Afebrile Patient
  * Without important electrolyte disorders

Exclusion Criteria:

* Obese patients with B.M.I. >35
* pregnant women
* patients <18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in the Intensive Care Unit of the University Hospital of Larissa
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2018-06-29 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
The correlation of inspiratory esophageal pressure, as assessed by esophageal manometry, to diaphragmatic thickness, as assessed by ultrasound, in patients who are weaned from mechanical ventilation. | 1 year
  The authors will study the correlation of inspiratory esophageal pressure, as assessed by esophageal manometry (values in cm H2O), to diaphragmatic thickness, as assessed by ultrasound (values in cm), in patients who are weaned from mechanical ventilation.Then a comparison will be made between the patients who failed and those who succeeded. Ten consecutive tidal breaths will be studied both by esophageal manometry and ultrasound of the diaphragm in each patient.

CONTACTS AND LOCATIONS:
Locations (1):
- Critical Care Unit, Larissa, Thessaly, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brochard L. (1991) Transdiaphragmatic Pressure. In: Benito S., Net A. (eds) Pulmonary Function in Mechanically Ventilated Patients. Update in Intensive Care and Emergency Medicine, vol 13. Springer, Berlin, Heidelberg
- [Background] Mauri T, Yoshida T, Bellani G, Goligher EC, Carteaux G, Rittayamai N, Mojoli F, Chiumello D, Piquilloud L, Grasso S, Jubran A, Laghi F, Magder S, Pesenti A, Loring S, Gattinoni L, Talmor D, Blanch L, Amato M, Chen L, Brochard L, Mancebo J; PLeUral pressure working Group (PLUG-Acute Respiratory Failure section of the European Society of Intensive Care Medicine). Esophageal and transpulmonary pressure in the clinical setting: meaning, usefulness and perspectives. Intensive Care Med. 2016 Sep;42(9):1360-73. doi: 10.1007/s00134-016-4400-x. Epub 2016 Jun 22. PMID 27334266
- [Background] Turnbull D, Webber S, Hamnegard CH, Mills GH. Intra-abdominal pressure measurement: validation of intragastric pressure as a measure of intra-abdominal pressure. Br J Anaesth. 2007 May;98(5):628-34. doi: 10.1093/bja/aem060. PMID 17456490
- [Background] Beaulieu Y, Marik PE. Bedside ultrasonography in the ICU: part 1. Chest. 2005 Aug;128(2):881-95. doi: 10.1378/chest.128.2.881. PMID 16100182
- [Background] Beaulieu Y, Marik PE. Bedside ultrasonography in the ICU: part 2. Chest. 2005 Sep;128(3):1766-81. doi: 10.1378/chest.128.3.1766. PMID 16162786
- [Background] Matamis D, Soilemezi E, Tsagourias M, Akoumianaki E, Dimassi S, Boroli F, Richard JC, Brochard L. Sonographic evaluation of the diaphragm in critically ill patients. Technique and clinical applications. Intensive Care Med. 2013 May;39(5):801-10. doi: 10.1007/s00134-013-2823-1. Epub 2013 Jan 24. PMID 23344830
- [Background] Goligher EC, Laghi F, Detsky ME, Farias P, Murray A, Brace D, Brochard LJ, Bolz SS, Rubenfeld GD, Kavanagh BP, Ferguson ND. Measuring diaphragm thickness with ultrasound in mechanically ventilated patients: feasibility, reproducibility and validity. Intensive Care Med. 2015 Apr;41(4):734. doi: 10.1007/s00134-015-3724-2. No abstract available. PMID 25749574
- [Background] MacIntyre NR, Cook DJ, Ely EW Jr, Epstein SK, Fink JB, Heffner JE, Hess D, Hubmayer RD, Scheinhorn DJ; American College of Chest Physicians; American Association for Respiratory Care; American College of Critical Care Medicine. Evidence-based guidelines for weaning and discontinuing ventilatory support: a collective task force facilitated by the American College of Chest Physicians; the American Association for Respiratory Care; and the American College of Critical Care Medicine. Chest. 2001 Dec;120(6 Suppl):375S-95S. doi: 10.1378/chest.120.6_suppl.375s. No abstract available. PMID 11742959
- [Background] MILIC-EMILI J, MEAD J, TURNER JM, GLAUSER EM. IMPROVED TECHNIQUE FOR ESTIMATING PLEURAL PRESSURE FROM ESOPHAGEAL BALLOONS. J Appl Physiol. 1964 Mar;19:207-11. doi: 10.1152/jappl.1964.19.2.207. No abstract available. PMID 14155283
- [Background] Baydur A, Behrakis PK, Zin WA, Jaeger M, Milic-Emili J. A simple method for assessing the validity of the esophageal balloon technique. Am Rev Respir Dis. 1982 Nov;126(5):788-91. doi: 10.1164/arrd.1982.126.5.788. PMID 7149443
- [Background] Bellemare F, Grassino A. Effect of pressure and timing of contraction on human diaphragm fatigue. J Appl Physiol Respir Environ Exerc Physiol. 1982 Nov;53(5):1190-5. doi: 10.1152/jappl.1982.53.5.1190. PMID 7174413
- [Background] Grinnan DC, Truwit JD. Clinical review: respiratory mechanics in spontaneous and assisted ventilation. Crit Care. 2005 Oct 5;9(5):472-84. doi: 10.1186/cc3516. Epub 2005 Apr 18. PMID 16277736
- [Background] Vivier E, Mekontso Dessap A, Dimassi S, Vargas F, Lyazidi A, Thille AW, Brochard L. Diaphragm ultrasonography to estimate the work of breathing during non-invasive ventilation. Intensive Care Med. 2012 May;38(5):796-803. doi: 10.1007/s00134-012-2547-7. Epub 2012 Apr 5. PMID 22476448
- [Background] Yang KL, Tobin MJ. A prospective study of indexes predicting the outcome of trials of weaning from mechanical ventilation. N Engl J Med. 1991 May 23;324(21):1445-50. doi: 10.1056/NEJM199105233242101. PMID 2023603
- [Background] Nemer SN, Barbas CS, Caldeira JB, Guimaraes B, Azeredo LM, Gago R, Souza PC. Evaluation of maximal inspiratory pressure, tracheal airway occlusion pressure, and its ratio in the weaning outcome. J Crit Care. 2009 Sep;24(3):441-6. doi: 10.1016/j.jcrc.2009.01.007. Epub 2009 Mar 27. PMID 19327955